CLINICAL TRIAL: NCT02271438
Title: A Randomized, Double-Blind, Placebo- and Positive-Controlled, Single-Dose, Four-Way Crossover Study to Evaluate the Effects of Ibrutinib on Cardiac Repolarization in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of Ibrutinib on Cardiac Repolarization in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR103807; PCI-32765CLL1007 (Other: Janssen Research & Development, LLC); 2014-000081-22 (EudraCT Number)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Healthy; Ibrutinib; Moxifloxacin; Cardiac Repolarization; Electrocardiogram; QTc interval
MeSH Terms: interventions — ibrutinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1: Ibrutinib 840 milligram (mg) (Experimental): Participants will receive ibrutinib 840 mg (6*140 mg capsules) + 6 placebo capsules on Day 1 of Part 1, Period 1.
  Interventions: Drug: Ibrutinib
- Part 1: Ibrutinib 1680 mg (Experimental): Participants will receive ibrutinib 1680 mg (12*140 mg capsules) on Day 1 of Part 1, Period 2.
  Interventions: Drug: Ibrutinib
- Part 2: Treatment A (Experimental): Participants will receive ibrutinib, 1680 mg (12*140 mg capsules) + 1 moxifloxacin-matching placebo capsule Day 1of Part 2.
  Interventions: Drug: Ibrutinib; Drug: Moxifloxacin-matching placebo
- Part 2: Treatment B (Experimental): Participants will receive ibrutinib, 840 mg (6*140 mg capsules) + 6 ibrutinib-matching placebo capsules + 1 moxifloxacin-matching placebo capsule.
  Interventions: Drug: Ibrutinib; Drug: Moxifloxacin-matching placebo
- Part 2: Treatment C (Experimental): Participants will receive placebo (12 ibrutinib-matching placebo capsules + 1 moxifloxacin-matching placebo capsule) Day 1 of Part 2.
  Interventions: Drug: Ibrutinib-matching placebo; Drug: Moxifloxacin-matching placebo
- Part 2: Treatment D (Experimental): Participants will receive moxifloxacin 400 mg (1 capsule) + 12 ibrutinib-matching placebo capsules Day 1 of Part 2.
  Interventions: Drug: Moxifloxacin; Drug: Ibrutinib-matching placebo

INTERVENTIONS:
Drug: Ibrutinib — Participants will receive a single oral dose of 12 capsules (12*140 mg capsules) of ibrutinib in Treatment A and 6 capsules (4 6*140 mg capsules) of ibrutinib in Treatment B.
  Arms: Part 1: Ibrutinib 1680 mg; Part 1: Ibrutinib 840 milligram (mg); Part 2: Treatment A; Part 2: Treatment B
Drug: Moxifloxacin — Participants will receive a single oral dose of 1 moxifloxacin capsule (400 mg) in Treatment D.
  Arms: Part 2: Treatment D
Drug: Ibrutinib-matching placebo — Participants will receive a single oral dose of 12 ibrutinib-matching placebo capsules in Treatment B and 6 ibrutinib-matching placebo capsules in Treatment C and D.
  Arms: Part 2: Treatment C; Part 2: Treatment D
Drug: Moxifloxacin-matching placebo — Participants will receive a single oral dose of 1 moxifloxacin-matching placebo capsule in Treatment A, B, and C.
  Arms: Part 2: Treatment A; Part 2: Treatment B; Part 2: Treatment C

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ibrutinib, to compare the pharmacokinetics of ibrutinib after single oral administration of 840 mg and 1680 mg and to assess the effects of a single dose of ibrutinib on QT/QTc intervals and electrocardiogram (ECG) in healthy adults.

DETAILED DESCRIPTION:
The study consists of 2 parts: Part 1 and Part 2. Part 1 is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving), single-center, 2-period, sequential design part. It consists of a Screening phase (Day-21 to -2), Treatment Period 1 and Treatment Period 2. In treatment period 1, 8 participants including two women will receive 840 milligram (mg) ibrutinib capsules + 6 placebo capsules. In treatment period 2, participants will receive 1680 mg ibrutinib capsules. Treatment periods will be separated by a Washout period of not less than 7 days. A high-fat breakfast will be provided 2 hours before dosing. Blood samples will be collected after each dosing for pharmacokinetic assessments.

Part 2 is a randomized (the study medication is assigned by chance), placebo (an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study) and positive-controlled (participants are assigned to either a recognized effective treatment or the study medication), double-blind (neither physician nor participant knows the treatment that the participant receives), single dose, and 4-way crossover (the same medications are provided to all participants but in a different sequence) part. Participants will receive either of the 4 treatments: Treatment A (Ibrutinib 1680 mg + moxifloxacin-matching placebo); Treatment B (Ibrutinib 840 mg+ ibrutinib-matching placebo + moxifloxacin-matching placebo); Treatment C (ibrutinib-matching placebo + moxifloxacin-matching placebo); and Treatment D: (moxifloxacin 400 mg + ibrutinib-matching placebo). Each treatment period will be separated by a Washout period of not less than 7 days. Electrocardiogram (ECG) will be recorded. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document indicating they understand the purpose of the study and procedures
* Must have a body mass index (BMI) of between 18 and 30 kg/m^2, inclusive
* Must have a body weight of not less than 50 kg
* Must have a blood pressure between 90 and 140 mmHg inclusive, systolic, and no higher than 90 mmHg diastolic at screening
* Must have an average of triplicate 12-lead ECG recordings, completed within 5 minutes total, consistent with normal cardiac conduction and function

Exclusion Criteria:

* History of or current clinically significant medical illness
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram
* History of clinically relevant heart rhythm disturbances including atrial, junctional, re-entry, and ventricular tachycardias, and heart blocks
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements
* Donated blood or blood products or had substantial loss of blood within 3 months before screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTc interval | Baseline (predose) up to Day 4
  The QTc interval, as measured by electrocardiograms will evaluate the potential effect of ibrutinib on QTc interval duration.
Number of Participants with Adverse events | Up to Day 12 of the follow-up period

SECONDARY OUTCOMES:
Change from baseline in RR interval | Baseline (predose) up to Day 4
  The RR interval is the portion between two consecutive R waves in the electrocardiogram.
Change from baseline in heart rate | Baseline (predose) up to Day 4
Change from baseline in PR interval | Baseline (predose) up to Day 4
  The PR interval is the portion of the electrocardiogram between the onset of the P wave (atrial depolarization) and the QRS complex (ventricular depolarization).
Change from baseline in QRS interval | Baseline (predose) up to Day 4
  The QRS interval is the interval from the beginning of the Q wave to the termination of the S wave, representing the time for ventricular depolarization.
Plasma concentration of ibrutinib following administration of a single dose | Predose (before tablet intake), up to 72 hours after dose
  Plasma concentrations of ibrutinib are used to evaluate when the highest concentration is achieved in the body and how long it stays in the body.
Plasma concentration of the Metabolite, PCI-45227, following administration of a single dose of ibrutinib | Predose (before tablet intake), up to 72 hours after dose
  Plasma concentrations of the metabolite, PCI-45227, are used to evaluate when the highest concentration is achieved in the body and how long it stays in the body.
Plasma concentration of moxifloxacin following administration of a single dose | Predose (before tablet intake), up to 72 hours after dose
  Plasma concentrations of moxifloxacin are used to evaluate when the highest concentration is achieved in the body and how long it stays in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] de Jong J, Hellemans P, Jiao JJ, Huang Y, Mesens S, Sukbuntherng J, Ouellet D. Ibrutinib does not prolong the corrected QT interval in healthy subjects: results from a thorough QT study. Cancer Chemother Pharmacol. 2017 Dec;80(6):1227-1237. doi: 10.1007/s00280-017-3471-x. Epub 2017 Oct 28. PMID 29080970